CLINICAL TRIAL: NCT02370992
Title: Prospective Multi-centre Study of Low-dose Rate Iodine125 (I-125) Prostate Brachytherapy Performed After Transurethral Resection
Brief Title: I125 Brachytherapy After TURP
Status: Completed | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CO11/9837
Record Dates: First submitted 2015-02-09; First posted 2015-02-25 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Receiving I125 brachytherapy: I125 brachytherapy is a standard treatment and will be delivered using routine techniques involving a preimplant volume study followed by implantation of the I125 sources. This is undertaken as an inpatient or day case under general or spinal anaesthetic according to local practice
  Interventions: Radiation: I125 brachytherapy

INTERVENTIONS:
Radiation: I125 brachytherapy — I125 brachytherapy is a standard treatment and will be delivered using routine techniques involving a preimplant volume study followed by implantation of the I125 sources. This is undertaken as an inpatient or day case under general or spinal anaesthetic according to local practice

SUMMARY:
Low dose rate brachytherapy using iodine 125 is well established as a treatment for low and intermediate risk prostate cancer. Currently there is uncertainty as to the safety of this technique in patients who have had a previous transurethral resection of the prostate gland (TURP) for obstruction of the urine flow through the prostatic urethra. Early experience when the technique was being developed in the 1980s suggested that there was a higher incidence of urinary incontinence after brachytherapy if there had been a previous TURP. It is however clear that with increasing experience many centres offer this treatment to patients who have had previous TURP, using various parameters to select patients including time from the TURP and persence or absence of a significant cavity within the gland on MRI scanning. There has been no systematic study of I125 brachytherapy after TURP in the current era which might address and inform the practice for future patient. Hence this study is designed to formally assess the safety of I125 brachytherapy after previous TURP.

ELIGIBILITY:
Inclusion Criteria:

* WHO performance status 0-1
* No contra-indication for anaesthesia
* No history of irradiation of the pelvis
* No other oncologic malignancy except adequately treated basal cell carcinoma of the skin or other malignancy from which the patient is disease free for at least 5 years.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule;

Prostate (cancer) related:

* Histologically proven prostate cancer (adenocarcinoma) of low or intermediate risk following the D'Amico classification.
* Prostate volume < 50 cc as measured on transrectal ultrasound
* Neo-adjuvant antiandrogen hormonal treatment is permitted to downsize the prostate volume or to cover waiting time till brachytherapy procedure. No adjuvant hormonal treatment is permitted.
* History of TransUrethral Resection of the prostate (TURp), performed at least 3 months before the brachytherapy procedure.
* Rim of prostate tissue of at least 1 cm around the post-TURp urethral defect at thepostero-lateral sides of the prostate
* Absence of significant TURp-induced urinary incontinence
* IPSS <15

Exclusion Criteria:

* Locally advanced (stage T3 or T4 , or metastatic (stage N+ or M+) prostate cancer High grade tumours defined by Gleason score 8 or above Co-morbidity which would exclude the patient from a transperineal implant procedure.

Unable to give informed consent.

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients taking part will do so having chosen I125 brachytherapy as their chosen treatment for prostate cancer and will have previously undergone TURP
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Change in acute and late urinary toxicity defined by International Prostate Specific Score and Common Terminology Criteria for Adverse Events v4. | Measured at 1 mth, 3 months, 6 month, 12 months, 18 months, 24 months and then yearly
  This change will be measured at 1 mth, 3 months, 6 month, 12 months, 18 months, 24 months and then yearly

SECONDARY OUTCOMES:
Gastro-intestinal and sexual function | Measured at 1 mth.
  Incidence of seed loss at 1 month and 6 months after implant and Biochemical disease free survival (Phoenix-definition.)
Gastro-intestinal and sexual function | Measured at 3 mth.
  Incidence of seed loss at 1 month and 6 months after implant and Biochemical disease free survival (Phoenix-definition.)
Gastro-intestinal and sexual function | Measured at 6 mth.
  Incidence of seed loss at 1 month and 6 months after implant and Biochemical disease free survival (Phoenix-definition.)
Gastro-intestinal and sexual function | Measured at 12 mth.
  Incidence of seed loss at 1 month and 6 months after implant and Biochemical disease free survival (Phoenix-definition.)

CONTACTS AND LOCATIONS:
Locations (1):
- The Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom